CLINICAL TRIAL: NCT06630871
Title: A Prospective, Multicenter, Single-Arm, Phase Ⅱ, Exploratory Clinical Trial Evaluating the Efficacy and Safety of Disitamab Vedotin Plus Tislelizumab Combined with Re-TURBT in the Treatment of HER-2-high Expression(2+-3+) Non-muscle Invasive Bladder Cancer At High-risk and Very High-risk.
Brief Title: A Clinical Trial Evaluating the Efficacy and Safety of Disitamab Vedotin Plus Tislelizumab Combined with Re-TURBT in the Treatment of HER-2-high Expression(2+-3+) Non-muscle Invasive Bladder Cancer At High-risk and Very High-risk.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: BeiGene (Industry); RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024YF042-01
Record Dates: First submitted 2024-09-25; First posted 2024-10-08 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: NMIBC
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): High risk and extremely high risk NMIBC for HER2 2 2+or 3+treated with combination therapy of trastuzumab, Distitamab Vedotin, and re-TURBt
  Interventions: Drug: Distitamab Vedotin in combination with Tislelizumab

INTERVENTIONS:
Drug: Distitamab Vedotin in combination with Tislelizumab — On the day after the initial TURBt procedure, use trastuzumab (200mg)+ Distitamab Vedotin (120mg [≤ 60Kg] or 2.0mg/Kg [>60Kg]) every 3 weeks (Q3W). Simultaneously arrange for the patient to complete a second TURBt within 6 weeks, and continue to use 3 courses of Trastuzumab+Vediximab (Q3W) after surgery until the endpoint of 3-year follow-up
  Other Names: surgery：re-TURBT

SUMMARY:
This prospective, multicenter, single-arm phase II trial aims to evaluate the clinical efficacy and safety of the combination therapy of Disitamab Vedotin with Tislelizumab and a second transurethral resection for the treatment of high-risk, very high-risk NMIBC with HER2 2+-3+.

DETAILED DESCRIPTION:
The specific implementation process of trial:

Patients diagnosed with high-risk and very high-risk NMIBC, based on medical history, clinical presentation, imaging examinations (such as MRI with plain and enhanced scanning), and transurethral resection for tissue pathological biopsy, are included in the "case screening process";. After excluding surgical contraindications, TURBt is performed; postoperative tissue pathological examination confirms NMIBC, and patients with immunohistochemical results of HER2 as 3+ or 2+ enter further screening. Referring to the AUA guidelines, high-risk and very high-risk NMIBC are included in subsequent analysis, where those who meet the inclusion criteria of this study, excluding the exclusion criteria, and who have recovered well after the initial TURBt and are assessed to be able to complete a second TURBt within six weeks are considered as the final candidates for enrollment.

Eligible patients for single-arm enrollment (N=40) will receive Tislelizumab (200mg) + Disitamab Vedotin (120mg for weight ≤60Kg or 2.0mg/Kg for weight ≥60Kg) the day after the initial TURBt, to be repeated every 3 weeks (Q3W). Patients are also scheduled to undergo a second TURBt within 6 weeks, and after the surgery, they will continue with three more courses of Tislelizumab + Disitamab Vedotin (Q3W) until the end of the 3-year follow-up period. The primary endpoint for evaluation in this study phase is the 1-year event-free survival (EFS), with secondary endpoints including 3-year EFS, 2-year bladder intact disease-free survival (BIDFS), time to total cystectomy, overall survival (OS), quality of life (QLQ-C30), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the experiment and sign a written informed consent form；
* Patients should be aged between 18 and 85 years, with no gender restrictions, no severe organ failure such as heart, lung, or brain, and an expected survival period of one year or more;
* Complete the relevant screening tests (routine blood test, coagulation function, liver and kidney function, infectious disease screening, 12-lead electrocardiogram, urinary system ultrasound, pelvic enhanced CT or MRI, and tissue pathology examination), and have no contraindications for TURBt surgery;
* Eastern Cooperative Oncology Group (ECOG) score: 0-2 points;
* Previous systemic therapy without systemic immunity/ADC drugs；
* Histologically confirmed non muscle invasive bladder cancer (NMIBC), with or without carcinoma in situ (CIS), the main pathological type is urothelial carcinoma, including other specific histopathological types, but urothelial carcinoma dominates (at least 50%). Patients with AUA classification of high-risk and extremely high-risk recurrence or progression risk by the American Urological Association, and with immunohistochemical results of Her2 being 3+or 2+, who have undergone maximal TURBt within 6 weeks.

Exclusion Criteria:

* Any of the following circumstances: those with immune deficiency or impairment (such as AIDS patients), who are using immunosuppressive drugs or radiotherapy, and who may cause systemic BCG disease reaction; Individuals who are allergic to the components of BCG vaccine; Patients with fever and acute infectious diseases, including active tuberculosis, or those receiving anti tuberculosis treatment; Accompanied by severe chronic cardiovascular and cerebrovascular diseases or chronic kidney disease;
* Patients with other urogenital system tumors or other organ tumors;
* Patients with AUA grading of low-risk, moderate risk NMIBC, or myometrial invasive bladder urothelial carcinoma (T2 stage or above), or immunohistochemistry Her2 negative or 1+patients;
* Individuals who have received chemotherapy, radiation therapy, or immunotherapy within the past 4 weeks;
* Pregnant or lactating women, women of childbearing age who have not taken effective contraceptive measures, and those planning to conceive during the trial period (including male subject partners);
* Patients with severe urethral stricture who cannot undergo cystoscopy, those with a history of bladder contracture or functional bladder volume less than 100mL;
* Patients with various mental disorders, severe coagulation function, liver and kidney function, hematopoietic dysfunction, etc. who cannot tolerate surgical treatment;
* Participated in clinical trials of other drugs within the past 3 months prior to enrollment;
* Known opioid or alcohol dependent individuals;
* Researchers believe that there may be any situation that increases the risk to participants or interferes with the execution of clinical trials.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
1-year Event-Free Survival rate | From date of randomization until the date of any event occurrence, whichever came first，assessed up to 12 months
  The possibility of patients have not experienced any events for at least 12 months after receiving treatment, including death, disease progression, switch to chemotherapy, addition of other treatments, fatal or intolerable side effects, etc

SECONDARY OUTCOMES:
3-years Event-Free Survival rate | From date of randomization until the date of any event occurrence, whichever came first，assessed up to 36 months
  The possibility of patients have not experienced any events for at least 36 months after receiving treatment, including death, disease progression, switch to chemotherapy, addition of other treatments, fatal or intolerable side effects, etc
2-year bladder disease-free survival（2 year BIDFS） rate | From date of randomization until the date of muscle-invasive recurrence, regional lymph node recurrence, distant metastasis, the need for radical cystectomy, or death, whichever came first，assessed up to 24 months
  The probability of patients remaining free from muscle-invasive recurrence, regional lymph node recurrence, distant metastasis, the need for radical cystectomy, or death for at least 24 months after the initiation of treatment
Reccurence Free Survival（ RFS） | From date of the first TURBT until the date of bladder tumor recurrence, assessed up to 36 months
  Time from the first TURBT to the first occurrence of bladder tumor recurrence was recorded by cystoscopy and pathological examination, with the main time points being 1 year, 2 years, and 3 years
Overall survival | From date of randomization until the date of death from any cause, assessed up to 60 months
  Time from the start of treatment to death from any causes
Time to complete bladder resection | From date of randomization until the date of radical cystectomy, assessed up to 60 months
  Time from the start of treatment to Radical cystectomy
Quality of life assessed by QLQ-C30 scale | through study completion, an average of 3 years
  Assessed by QLQ-C30 scale, higher scores mean better outcomes
Adverse events | through study completion, an average of 3 years
  The type, incidence, relatedness, and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No